CLINICAL TRIAL: NCT01307501
Title: Evaluating Cryoablation of Metastatic Lung/Pleura Tumors in Patients - Safety and Efficacy
Brief Title: Safety and Efficacy of Cryoablation for Metastatic Lung Tumors
Acronym: ECLIPSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CUC10-LNG06
Record Dates: First submitted 2011-03-01; First posted 2011-03-03 (Estimated); Results first posted 2019-10-01 (Actual); Last update posted 2021-07-19 (Actual); Status verified 2021-07

CONDITIONS: Metastatic Lung Cancer
Keywords: Cryoablation; Cryotherapy; Cryosurgery; Metastatic; Lung; Pleura; Tumors
MeSH Terms: conditions — Lung Neoplasms; Neoplasm Metastasis; Neoplasms | interventions — Cryosurgery

STUDY DESIGN:
Intervention Model Description: All participants received the same treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Cryoablation (Other): Participants will undergo a cryoablation procedure with the Galil Medical Cryoablation System according to the manufacturer's guidelines. Participant preparation, anesthesia, intra-operative monitoring, and postoperative management for the study cryoablation procedure will be identical to those for standard cryoablation treatment routinely performed at the clinical centers that participated in this study and will be at the discretion of the Investigators. No more than 3 tumors in 1 lung can be treated in a single session, and no more than 5 total lung tumors (across both lungs) can be treated during the study.
  Interventions: Device: Cryoablation

INTERVENTIONS:
Device: Cryoablation — Application of extremely cold temperatures to the identified tumor(s).
  Other Names: Visual-ICE® Cryoablation System; PresIce® Cryoablation System; SeedNet® Cryoablation System; IceRod® Cryoablation Needles; IceRod® PLUS Cryoablation Needles; IceSphere™ Cryoablation Needles; IceSeed™ Cryoablation Needles; IceEDGE™ 2.4 Cryoablation Needles

SUMMARY:
ECLIPSE will evaluate the safety and efficacy of cryoablation therapy used to treat tumors less than or equal to 3.5 centimeters (cm) in participants with pulmonary metastatic disease.

DETAILED DESCRIPTION:
ECLIPSE is a treatment, Phase 1 multicenter, prospective, single-arm study with participants serving as their own control. This study is to enroll participants who will undergo cryoablation of at least 1 metastatic pulmonary tumor that is less than or equal to 3.5 cm. Participants will be followed for 5 years post their cryoablation procedure.

Cryoablation is the process of destroying tissue by the application of extremely cold temperatures. Galil Medical Cryoablation Systems are used as a surgical tool in the fields of general surgery, dermatology (skin), neurology (nerves), chest surgery (including lung), Ears-Nose-Throat (ENT), gynecology, oncology (cancer), proctology (colon/rectal), and urology (kidney).

ELIGIBILITY:
Inclusion Criteria:

* Participant must be at least 18 years old.
* Participant has signed a written informed consent.
* Participant presents with Stage 4 pulmonary metastatic disease with metastatic disease previously confirmed by prior biopsy or confirmed on imaging with known primary disease.
* Participant has up to 3 local metastases unilaterally targeted by cryoablation. Maximum of 5 total pulmonary tumors bilaterally.
* Targeted tumor(s) defined as intra pulmonary or pleural with a maximum size of 3.5 cm.
* The target tumor is determined (by CT/MRI) to be in a location where cryoablation is technically achievable based on the proximity of adjacent organs and structures.
* Eastern Cooperative Oncology Group (ECOG) score of 0-2.
* Karnofsky Performance Scale (KPS) score ≥60.
* Platelet count >50,000/cubed millimeters (mm^3) within 60 days prior to study treatment.
* International normalized ratio (INR) less than 1.5 within 60 days prior to study treatment.
* Participant has a life expectancy of >3 months.
* Participant is clinically suitable for cryoablation procedure.

Exclusion Criteria:

* Participant's primary cancer is lung cancer.
* Participant is unable to lie flat or has respiratory distress at rest.
* Participant has uncontrolled coagulopathy or bleeding disorders.
* Participant has had chemotherapy with neutropenia to levels as confirmed by absolute neutrophil count (ANC) of less than 1000 that produce increase risk for the cryoablation procedure.
* Participant has a history of an allergic reaction to iodine injections or to shellfish.
* Participant has evidence of active systemic, pulmonary, or pericardial infection.
* Participant has a debilitating medical or psychiatric illness that would preclude giving informed consent or receiving optimal treatment or follow up.
* Participant is currently participating in other experimental studies that could affect the primary endpoint.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-01-04 (Actual); Primary Completion 2018-08-30 (Actual); Study Completion 2018-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hiran Fernando, MD, Study Chair — Boston Medical Center
Locations (4):
- United States (3):
  - Ronald Regan UCLA Medical Center, Los Angeles, California
  - Karmanos Cancer Institute, Detroit, Michigan
  - Mayo Clinic Rochester, Rochester, Minnesota
- Institut Gustave Roussy, Villejuif, Cedex, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gillams A. Lung tumour ablation - where are we now? Cancer Imaging. 2008 Apr 22;8(1):116-7. doi: 10.1102/1470-7330.2008.0015. PMID 18442957
- [Background] Ahmed A, Littrup P. Percutaneous cryotherapy of the thorax: safety considerations for complex cases. AJR Am J Roentgenol. 2006 Jun;186(6):1703-6. doi: 10.2214/AJR.04.1068. No abstract available. PMID 16714662
- [Background] Asimakopoulos G, Beeson J, Evans J, Maiwand MO. Cryosurgery for malignant endobronchial tumors: analysis of outcome. Chest. 2005 Jun;127(6):2007-14. doi: 10.1378/chest.127.6.2007. PMID 15947313
- [Background] Kawamura M, Izumi Y, Tsukada N, Asakura K, Sugiura H, Yashiro H, Nakano K, Nakatsuka S, Kuribayashi S, Kobayashi K. Percutaneous cryoablation of small pulmonary malignant tumors under computed tomographic guidance with local anesthesia for nonsurgical candidates. J Thorac Cardiovasc Surg. 2006 May;131(5):1007-13. doi: 10.1016/j.jtcvs.2005.12.051. PMID 16678583
- [Background] Wang H, Littrup PJ, Duan Y, Zhang Y, Feng H, Nie Z. Thoracic masses treated with percutaneous cryotherapy: initial experience with more than 200 procedures. Radiology. 2005 Apr;235(1):289-98. doi: 10.1148/radiol.2351030747. PMID 15798173
- [Background] Blazeby JM, Avery K, Sprangers M, Pikhart H, Fayers P, Donovan J. Health-related quality of life measurement in randomized clinical trials in surgical oncology. J Clin Oncol. 2006 Jul 1;24(19):3178-86. doi: 10.1200/JCO.2005.05.2951. PMID 16809741
- [Background] Ware J Jr, Kosinski M, Keller SD. A 12-Item Short-Form Health Survey: construction of scales and preliminary tests of reliability and validity. Med Care. 1996 Mar;34(3):220-33. doi: 10.1097/00005650-199603000-00003. PMID 8628042

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Index Tumors
Groups:
- Cryoablation: Participants underwent a cryoablation procedure with the Galil Medical Cryoablation System according to the manufacturer's guidelines. Participant preparation, anesthesia, intra-operative monitoring, and postoperative management for the study cryoablation procedure were identical to those for standard cryoablation treatment routinely performed at the clinical centers that participated in this study and were at the discretion of the Investigators. No more than 3 tumors in 1 lung were treated in a single session, and no more than 5 total lung tumors (across both lungs) were treated during the study.
Period: Overall Study
Arm/Group | Cryoablation
Started | 40; 60 Index Tumors
Intent-to-Treat (ITT) Population (Participants for whom cryoablation via Galil Medical Cryoablation System was attempted or performed.) | 40; 60 Index Tumors
Completed | 17; 23 Index Tumors
Not Completed | 23; 37 Index Tumors
Not completed — Treatment Failure | 1
Not completed — Death | 20
Not completed — Lost to Follow-up | 1
Not completed — Starting Hospice | 1

BASELINE CHARACTERISTICS:
Population: Participants for whom cryoablation via Galil Medical Cryoablation System was attempted or performed (ITT Population).
Arm/Group | Cryoablation
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.6 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 17
  More than one race | 1
  Unknown or Not Reported | 19
Eastern Cooperative Oncology Group (ECOG) Performance Status [Mean (Standard Deviation); unit: score on a scale] — ECOG Performance Status Scoring: 0=Fully active, able to carry on all pre-disease performance without restriction; 1=Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature (for example, light house work, office work); 2=Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours; 3=Capable of only limited self-care, confined to bed or chair more than 50% of waking hours; 4=Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair; 5=Dead.
  score on a scale | 0.3 (0.5)
Physical Function as Assessed by the Karnofsky Performance Status (KPS) Scale [Mean (Standard Deviation); unit: score on a scale] — The KPS Scale is a standard way of measuring the ability of cancer patients to perform ordinary tasks. The scores range from 0 to 100. A higher score means the participant is better able to carry out daily activities. KPS may be used to determine a participant's prognosis, to measure changes in a participant's ability to function.
  score on a scale | 95.5 (8.1)
Quality of Life Over Time as Assessed by the Short Form-12 (SF-12) Generic Measure [Mean (Standard Deviation); unit: score on a scale] — The SF-12 is a shortened version of the well-known SF-36. The SF-12 assesses eight domains (physical functioning, role limitations due to physical health problems, bodily pain, social functioning, general mental health, role limitations due to emotional problems, vitality and general health perception). Assessments were made by examining the change in the baseline scores to those reported post-operatively. The scores range from 0 to 100. A higher value indicates a better quality of life of the participant.
  score on a scale
    Physical Functioning | 71.2 (34.9)
    Role Physical | 62.1 (29.7)
    Bodily Pain | 77.3 (26.8)
    Social Functioning | 80.5 (26.7)
    Mental Health | 69.5 (18.2)
    Role Emotional | 78.4 (21.0)
    Vitality | 57.8 (22.4)
    General Health Perception | 63.9 (23.3)

OUTCOME MEASURES:

1. Primary Outcome: Local Tumor Control for Each Index Tumor as Measured by Imaging at Month 60
Description: Local tumor control was achieved if either the greatest trans-axial diameter of a treated tumor was ≤20% greater than at the pre-procedure assessment (per-tumor assessment) or if the sum of greatest trans-axial diameters of all treated tumors for a participant was ≤20% greater than the sum for the pre-procedure assessment of those tumors (per-participant assessment). Complete Response defined as tumor disappearance (scar) or <25% of original size. If tumor/ablation zone had likely disappeared, the measurement was recorded as 0 mm; if tumor/ablation zone was present but too small to measure, the measurement was recorded as 5 mm. Partial Response defined as greater than 30% decrease in sum of the largest diameter of all targeted tumors. Stable Disease defined as less than 30% decrease in sum of the largest diameter of all targeted tumors. Local Failure defined as greater than 20% increase in the sum of the largest diameter of all targeted tumors. Worst response per participant was used.
Time Frame: Baseline and Month 60
Population: Participants for whom cryoablation via Galil Medical Cryoablation System was attempted or performed (ITT Population) with available data at the respective time point.
Measure: Number (95% Confidence Interval); unit: percentage of tumors
Units Other Than Participants: Tumors
Arm/Group | Cryoablation
Number analyzed (Participants) | 40
Number analyzed (Tumors) | 60
percentage of tumors
  Local Control, Month 60: number analyzed (Participants) | 16
  Local Control, Month 60: number analyzed (Tumors) | 20
  Local Control, Month 60 | 80.0 [56.3 to 94.3]
  Complete Response, Month 60: number analyzed (Participants) | 16
  Complete Response, Month 60: number analyzed (Tumors) | 20
  Complete Response, Month 60 | 45.0 [23.1 to 68.5]
  Partial Response, Month 60: number analyzed (Participants) | 16
  Partial Response, Month 60: number analyzed (Tumors) | 20
  Partial Response, Month 60 | 15.0 [3.2 to 37.9]
  Stable Disease, Month 60: number analyzed (Participants) | 16
  Stable Disease, Month 60: number analyzed (Tumors) | 20
  Stable Disease, Month 60 | 20.0 [5.7 to 43.7]
  Local Failure, Month 60: number analyzed (Participants) | 16
  Local Failure, Month 60: number analyzed (Tumors) | 20
  Local Failure, Month 60 | 20.0 [5.7 to 43.7]

2. Secondary Outcome: Local Tumor Control for Each Index Tumor as Measured by Imaging at Months 3, 6, 12, 24, 36, and 48
Description: Local tumor control was achieved if the greatest trans-axial diameter of a treated tumor was ≤20% greater than at the pre-procedure assessment (per-tumor assessment) or if the sum of the greatest trans-axial diameters of all treated tumors for a participant was ≤20% greater than the sum for the pre-procedure assessment of those tumors (per-participant assessment). Complete Response defined as tumor disappearance (scar) or <25% of original size. If tumor/ablation zone had likely disappeared, the measurement was recorded as 0 mm; if tumor/ablation zone was present but too small to measure, the measurement was recorded as 5 mm. Partial Response defined as greater than 30% decrease in sum of the largest diameter of all targeted tumors. Stable Disease defined as less than 30% decrease in sum of the largest diameter of all targeted tumors. Local Failure defined as greater than 20% increase in the sum of the largest diameter of all targeted tumors. Worst response per participant was used.
Time Frame: Baseline and Months 3, 6, 12, 24, 36, and 48
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of tumors
Units Other Than Participants: Tumors
Arm/Group | Cryoablation
Number analyzed (Participants) | 40
Number analyzed (Tumors) | 60
percentage of tumors
  Local Control, Month 3: number analyzed (Participants) | 37
  Local Control, Month 3: number analyzed (Tumors) | 56
  Local Control, Month 3 | 46.4 [33.0 to 60.3]
  Local Control, Month 6: number analyzed (Participants) | 37
  Local Control, Month 6: number analyzed (Tumors) | 57
  Local Control, Month 6 | 66.7 [52.9 to 78.6]
  Local Control, Month 12: number analyzed (Participants) | 34
  Local Control, Month 12: number analyzed (Tumors) | 51
  Local Control, Month 12 | 80.4 [66.9 to 90.2]
  Local Control, Month 24: number analyzed (Participants) | 27
  Local Control, Month 24: number analyzed (Tumors) | 40
  Local Control, Month 24 | 87.5 [73.2 to 95.8]
  Local Control, Month 48: number analyzed (Participants) | 19
  Local Control, Month 48: number analyzed (Tumors) | 22
  Local Control, Month 48 | 90.9 [70.8 to 98.9]
  Local Control, Month 36: number analyzed (Participants) | 23
  Local Control, Month 36: number analyzed (Tumors) | 31
  Local Control, Month 36 | 90.3 [74.2 to 98.0]
  Complete Response, Month 3: number analyzed (Participants) | 37
  Complete Response, Month 3: number analyzed (Tumors) | 56
  Complete Response, Month 3 | 5.4 [1.1 to 14.9]
  Complete Response, Month 6: number analyzed (Participants) | 37
  Complete Response, Month 6: number analyzed (Tumors) | 57
  Complete Response, Month 6 | 15.8 [7.5 to 27.9]
  Complete Response, Month 12: number analyzed (Participants) | 34
  Complete Response, Month 12: number analyzed (Tumors) | 51
  Complete Response, Month 12 | 23.5 [12.8 to 37.5]
  Complete Response, Month 24: number analyzed (Participants) | 27
  Complete Response, Month 24: number analyzed (Tumors) | 40
  Complete Response, Month 24 | 40.0 [24.9 to 56.7]
  Complete Response, Month 36: number analyzed (Participants) | 23
  Complete Response, Month 36: number analyzed (Tumors) | 31
  Complete Response, Month 36 | 38.7 [21.8 to 57.8]
  Complete Response, Month 48: number analyzed (Participants) | 19
  Complete Response, Month 48: number analyzed (Tumors) | 22
  Complete Response, Month 48 | 40.9 [20.7 to 63.6]
  Partial Response, Month 3: number analyzed (Participants) | 37
  Partial Response, Month 3: number analyzed (Tumors) | 56
  Partial Response, Month 3 | 3.6 [0.4 to 12.3]
  Partial Response, Month 6: number analyzed (Participants) | 37
  Partial Response, Month 6: number analyzed (Tumors) | 57
  Partial Response, Month 6 | 10.5 [4.0 to 21.5]
  Partial Response, Month 12: number analyzed (Participants) | 34
  Partial Response, Month 12: number analyzed (Tumors) | 51
  Partial Response, Month 12 | 15.7 [7.0 to 28.6]
  Partial Response, Month 24: number analyzed (Participants) | 27
  Partial Response, Month 24: number analyzed (Tumors) | 40
  Partial Response, Month 24 | 10.0 [2.8 to 23.7]
  Partial Response, Month 36: number analyzed (Participants) | 23
  Partial Response, Month 36: number analyzed (Tumors) | 31
  Partial Response, Month 36 | 16.1 [5.5 to 33.7]
  Partial Response, Month 48: number analyzed (Participants) | 19
  Partial Response, Month 48: number analyzed (Tumors) | 22
  Partial Response, Month 48 | 22.7 [7.8 to 45.4]
  Stable Disease, Month 3: number analyzed (Participants) | 37
  Stable Disease, Month 3: number analyzed (Tumors) | 56
  Stable Disease, Month 3 | 37.5 [24.9 to 51.5]
  Stable Disease, Month 6: number analyzed (Participants) | 37
  Stable Disease, Month 6: number analyzed (Tumors) | 57
  Stable Disease, Month 6 | 40.4 [27.6 to 54.2]
  Stable Disease, Month 12: number analyzed (Participants) | 34
  Stable Disease, Month 12: number analyzed (Tumors) | 51
  Stable Disease, Month 12 | 41.2 [27.6 to 55.8]
  Stable Disease, Month 24: number analyzed (Participants) | 27
  Stable Disease, Month 24: number analyzed (Tumors) | 40
  Stable Disease, Month 24 | 37.5 [22.7 to 54.2]
  Stable Disease, Month 36: number analyzed (Participants) | 23
  Stable Disease, Month 36: number analyzed (Tumors) | 31
  Stable Disease, Month 36 | 35.5 [19.2 to 54.6]
  Stable Disease, Month 48: number analyzed (Participants) | 19
  Stable Disease, Month 48: number analyzed (Tumors) | 22
  Stable Disease, Month 48 | 27.3 [10.7 to 50.2]
  Local Failure, Month 3: number analyzed (Participants) | 37
  Local Failure, Month 3: number analyzed (Tumors) | 56
  Local Failure, Month 3 | 53.6 [39.7 to 67.0]
  Local Failure, Month 6: number analyzed (Participants) | 37
  Local Failure, Month 6: number analyzed (Tumors) | 57
  Local Failure, Month 6 | 33.3 [21.4 to 47.1]
  Local Failure, Month 12: number analyzed (Participants) | 34
  Local Failure, Month 12: number analyzed (Tumors) | 51
  Local Failure, Month 12 | 19.6 [9.8 to 33.1]
  Local Failure, Month 24: number analyzed (Participants) | 27
  Local Failure, Month 24: number analyzed (Tumors) | 40
  Local Failure, Month 24 | 12.5 [4.2 to 26.8]
  Local Failure, Month 36: number analyzed (Participants) | 23
  Local Failure, Month 36: number analyzed (Tumors) | 31
  Local Failure, Month 36 | 9.7 [2.0 to 25.8]
  Local Failure, Month 48: number analyzed (Participants) | 19
  Local Failure, Month 48: number analyzed (Tumors) | 22
  Local Failure, Month 48 | 9.1 [1.1 to 29.2]

3. Secondary Outcome: Overall Disease-Specific Participant Survival Post-Cryoablation
Description: Disease-specific survival was analyzed as time in days from study cryoablation to participant death due to lung cancer. All deaths with documented lung disease progression were categorized as disease-specific deaths for this analysis. Participants who were alive were censored at the date of their last visit. Participants who died from causes other than lung cancer and did not have documented disease progression were censored at the time of death.
Time Frame: Up to Month 60
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Cryoablation
Number analyzed (Participants) | 40
percentage of participants
  Week 1 | 100
  Month 1 | 100
  Month 3 | 100
  Month 6: number analyzed (Participants) | 39
  Month 6 | 100
  Month 12: number analyzed (Participants) | 38
  Month 12 | 100
  Month 24: number analyzed (Participants) | 32
  Month 24 | 86.5
  Month 36: number analyzed (Participants) | 24
  Month 36 | 74.8
  Month 48: number analyzed (Participants) | 22
  Month 48 | 71.5
  Month 60: number analyzed (Participants) | 7
  Month 60 | 55.3

4. Secondary Outcome: Time in Days to Disease Recurrence or Progression Following Study Cryoablation
Description: Disease recurrence or progression will be determined locally by evidence of an increase in tumor size and/or contrast enhancement that met the definition of local tumor failure. Local tumor failure defined as a >20% increase from baseline in the sum of the largest diameter of all targeted tumors. Participants without disease recurrence or progression were censored at the date of their last visit or their date of death due to any cause. The percentage of participants with disease recurrence or progression after the study cryoablation procedure at the specified number of days is presented.
Time Frame: Baseline (0 days), Week 1 (7 days), and Months 3 (90 days), 6 (180 days), 12 (365 days), 24 (730 days), 36 (1095 days), 48 (1460 days), and 60 (1825 days)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Cryoablation
Number analyzed (Participants) | 40
percentage of participants
  Baseline | 0
  Week 1 (7 days) | 0
  Month 1 (30 days) | 0
  Month 3 (90 days) | 0
  Month 6 (180 days): number analyzed (Participants) | 38
  Month 6 (180 days) | 2.5
  Month 12 (365 days): number analyzed (Participants) | 37
  Month 12 (365 days) | 5.1
  Month 24 (730 days): number analyzed (Participants) | 30
  Month 24 (730 days) | 10.7
  Month 36 (1095 days): number analyzed (Participants) | 23
  Month 36 (1095 days) | 10.7
  Month 48 (1460 days): number analyzed (Participants) | 21
  Month 48 (1460 days) | 10.7
  Month 60 (1825 days): number analyzed (Participants) | 7
  Month 60 (1825 days) | 21.8

5. Secondary Outcome: Change From Baseline in ECOG Performance Status at Week 1 and Months 3, 6, 12, 24, 36, 48, and 60
Description: ECOG Performance Status defined as a set of criteria with corresponding scores used by the Investigator to assess how a participant's disease is progressing, assess how the disease affects the daily living abilities of the participant, and determine appropriate treatment and prognosis. ECOG Performance Status Scoring: 0=Fully active, able to carry on all pre-disease performance without restriction; 1=Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature (for example, light house work, office work); 2=Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours; 3=Capable of only limited self-care, confined to bed or chair more than 50% of waking hours; 4=Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair; 5=Dead.
Time Frame: Baseline, Week 1 and Months 3, 6, 12, 24, 36, 48, and 60
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cryoablation
Number analyzed (Participants) | 40
score on a scale
  Change at Week 1: number analyzed (Participants) | 38
  Change at Week 1 | 0.1 (0.5)
  Change at Month 1: number analyzed (Participants) | 22
  Change at Month 1 | 0 (0.4)
  Change at Month 3: number analyzed (Participants) | 32
  Change at Month 3 | 0.2 (0.4)
  Change at Month 6: number analyzed (Participants) | 31
  Change at Month 6 | 0.1 (0.4)
  Change at Month 12: number analyzed (Participants) | 27
  Change at Month 12 | 0.2 (0.6)
  Change at Month 24: number analyzed (Participants) | 20
  Change at Month 24 | 0.2 (0.6)
  Change at Month 36: number analyzed (Participants) | 15
  Change at Month 36 | -0.1 (0.5)
  Change at Month 48: number analyzed (Participants) | 14
  Change at Month 48 | 0.2 (0.8)
  Change at Month 60: number analyzed (Participants) | 12
  Change at Month 60 | 0.6 (1.0)

6. Secondary Outcome: Change From Baseline in Physical Function as Assessed by the KPS Scale at Week 1 and Months 3, 6, 12, 24, 36, 48, and 60
Description: The KPS Scale is a standard way of measuring the ability of cancer patients to perform ordinary tasks. The scores range from 0 to 100. A higher score means the participant is better able to carry out daily activities. KPS may be used to determine a participant's prognosis, to measure changes in a participant's ability to function.
Time Frame: Baseline, Week 1 and Months 3, 6, 12, 24, 36, 48, and 60
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cryoablation
Number analyzed (Participants) | 40
score on a scale
  Baseline | 95.5 (8.1)
  Change at Week 1: number analyzed (Participants) | 38
  Change at Week 1 | -1.8 (6.1)
  Change at Month 1: number analyzed (Participants) | 22
  Change at Month 1 | -0.9 (5.3)
  Change at Month 3: number analyzed (Participants) | 32
  Change at Month 3 | -1.6 (6.3)
  Change at Month 6: number analyzed (Participants) | 30
  Change at Month 6 | 0.3 (7.2)
  Change at Month 12: number analyzed (Participants) | 22
  Change at Month 12 | -0.5 (8.4)
  Change at Month 24: number analyzed (Participants) | 9
  Change at Month 24 | 4.4 (7.3)
  Change at Month 36: number analyzed (Participants) | 9
  Change at Month 36 | 7.8 (4.4)
  Change at Month 48: number analyzed (Participants) | 6
  Change at Month 48 | 5.0 (5.5)
  Change at Month 60: number analyzed (Participants) | 3
  Change at Month 60 | 6.7 (5.8)

7. Secondary Outcome: Change From Baseline in Quality of Life Over Time as Assessed by the SF-12 Generic Measure at Months 1, 3, 6, 12, 24, 36, 48, and 60
Description: The SF-12 is a shortened version of the well-known SF-36. The SF-12 assesses eight domains (physical functioning, role limitations due to physical health problems, bodily pain, social functioning, general mental health, role limitations due to emotional problems, vitality and general health perception). Assessments were made by examining the change in the baseline scores to those reported post-operatively. The scores range from 0 to 100. A higher value indicates a better quality of life of the participant.
Time Frame: Baseline, Months 1, 3, 6, 12, 24, 36, 48, and 60
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cryoablation
Number analyzed (Participants) | 40
score on a scale
  Physical Functioning, Change at Month 1: number analyzed (Participants) | 30
  Physical Functioning, Change at Month 1 | -10.0 (24.2)
  Physical Functioning, Change at Month 3: number analyzed (Participants) | 27
  Physical Functioning, Change at Month 3 | -12.0 (24.4)
  Physical Functioning, Change at Month 6: number analyzed (Participants) | 28
  Physical Functioning, Change at Month 6 | -12.5 (33.0)
  Physical Functioning, Change at Month 12: number analyzed (Participants) | 23
  Physical Functioning, Change at Month 12 | -23.9 (38.0)
  Physical Functioning, Change at Month 24: number analyzed (Participants) | 12
  Physical Functioning, Change at Month 24 | -10.4 (44.5)
  Physical Functioning, Change at Month 36: number analyzed (Participants) | 10
  Physical Functioning, Change at Month 36 | -12.5 (31.7)
  Physical Functioning, Change at Month 48: number analyzed (Participants) | 7
  Physical Functioning, Change at Month 48 | -10.7 (31.8)
  Physical Functioning, Change at Month 60: number analyzed (Participants) | 6
  Physical Functioning, Change at Month 60 | -12.5 (54.2)
  Role Physical, Change at Month 1: number analyzed (Participants) | 30
  Role Physical, Change at Month 1 | 4.2 (24.2)
  Role Physical, Change at Month 3: number analyzed (Participants) | 27
  Role Physical, Change at Month 3 | -1.9 (21.0)
  Role Physical, Change at Month 6: number analyzed (Participants) | 28
  Role Physical, Change at Month 6 | -0.4 (19.7)
  Role Physical, Change at Month 12: number analyzed (Participants) | 23
  Role Physical, Change at Month 12 | -2.2 (26.8)
  Role Physical, Change at Month 24: number analyzed (Participants) | 12
  Role Physical, Change at Month 24 | 5.2 (23.5)
  Role Physical, Change at Month 36: number analyzed (Participants) | 10
  Role Physical, Change at Month 36 | 5.0 (25.8)
  Role Physical, Change at Month 48: number analyzed (Participants) | 7
  Role Physical, Change at Month 48 | 3.6 (35.9)
  Role Physical, Change at Month 60: number analyzed (Participants) | 6
  Role Physical, Change at Month 60 | -4.2 (25.8)
  Bodily Pain, Change at Month 1: number analyzed (Participants) | 30
  Bodily Pain, Change at Month 1 | -9.2 (25.8)
  Bodily Pain, Change at Month 3: number analyzed (Participants) | 27
  Bodily Pain, Change at Month 3 | -3.7 (21.6)
  Bodily Pain, Change at Month 6: number analyzed (Participants) | 28
  Bodily Pain, Change at Month 6 | -9.8 (24.9)
  Bodily Pain, Change at Month 12: number analyzed (Participants) | 23
  Bodily Pain, Change at Month 12 | -7.6 (19.1)
  Bodily Pain, Change at Month 24: number analyzed (Participants) | 12
  Bodily Pain, Change at Month 24 | -18.8 (32.2)
  Bodily Pain, Change at Month 36: number analyzed (Participants) | 10
  Bodily Pain, Change at Month 36 | -5.0 (30.7)
  Bodily Pain, Change at Month 48: number analyzed (Participants) | 7
  Bodily Pain, Change at Month 48 | 0 (28.9)
  Bodily Pain, Change at Month 60: number analyzed (Participants) | 6
  Bodily Pain, Change at Month 60 | -8.3 (49.2)
  Social Functioning, Change at Month 1: number analyzed (Participants) | 29
  Social Functioning, Change at Month 1 | -8.6 (26.1)
  Social Functioning, Change at Month 3: number analyzed (Participants) | 27
  Social Functioning, Change at Month 3 | -3.7 (23.7)
  Social Functioning, Change at Month 6: number analyzed (Participants) | 27
  Social Functioning, Change at Month 6 | -4.6 (22.0)
  Social Functioning, Change at Month 12: number analyzed (Participants) | 22
  Social Functioning, Change at Month 12 | -11.4 (24.1)
  Social Functioning, Change at Month 24: number analyzed (Participants) | 12
  Social Functioning, Change at Month 24 | -12.5 (32.9)
  Social Functioning, Change at Month 36: number analyzed (Participants) | 10
  Social Functioning, Change at Month 36 | -2.5 (24.9)
  Social Functioning, Change at Month 48: number analyzed (Participants) | 7
  Social Functioning, Change at Month 48 | -3.6 (39.3)
  Social Functioning, Change at Month 60: number analyzed (Participants) | 6
  Social Functioning, Change at Month 60 | -12.5 (37.9)
  Mental Health, Change at Month 1: number analyzed (Participants) | 29
  Mental Health, Change at Month 1 | 1.7 (16.3)
  Mental Health, Change at Month 3: number analyzed (Participants) | 27
  Mental Health, Change at Month 3 | 0.9 (12.0)
  Mental Health, Change at Month 6: number analyzed (Participants) | 27
  Mental Health, Change at Month 6 | -1.4 (10.6)
  Mental Health, Change at Month 12: number analyzed (Participants) | 22
  Mental Health, Change at Month 12 | -0.6 (20.6)
  Mental Health, Change at Month 24: number analyzed (Participants) | 12
  Mental Health, Change at Month 24 | -3.1 (17.0)
  Mental Health, Change at Month 36: number analyzed (Participants) | 10
  Mental Health, Change at Month 36 | 3.8 (15.6)
  Mental Health, Change at Month 48: number analyzed (Participants) | 7
  Mental Health, Change at Month 48 | 8.9 (9.4)
  Mental Health, Change at Month 60: number analyzed (Participants) | 6
  Mental Health, Change at Month 60 | 0 (13.7)
  Role Emotional, Change at Month 1: number analyzed (Participants) | 30
  Role Emotional, Change at Month 1 | -3.3 (20.5)
  Role Emotional, Change at Month 3: number analyzed (Participants) | 27
  Role Emotional, Change at Month 3 | -11.6 (23.0)
  Role Emotional, Change at Month 6: number analyzed (Participants) | 28
  Role Emotional, Change at Month 6 | -2.7 (24.4)
  Role Emotional, Change at Month 12: number analyzed (Participants) | 23
  Role Emotional, Change at Month 12 | -3.8 (21.1)
  Role Emotional, Change at Month 24: number analyzed (Participants) | 12
  Role Emotional, Change at Month 24 | -11.5 (24.1)
  Role Emotional, Change at Month 36: number analyzed (Participants) | 10
  Role Emotional, Change at Month 36 | -11.3 (27.9)
  Role Emotional, Change at Month 48: number analyzed (Participants) | 7
  Role Emotional, Change at Month 48 | -8.9 (15.7)
  Role Emotional, Change at Month 60: number analyzed (Participants) | 6
  Role Emotional, Change at Month 60 | -22.9 (26.7)
  Vitality, Change at Month 1: number analyzed (Participants) | 29
  Vitality, Change at Month 1 | -6.0 (22.8)
  Vitality, Change at Month 3: number analyzed (Participants) | 27
  Vitality, Change at Month 3 | -9.3 (19.8)
  Vitality, Change at Month 6: number analyzed (Participants) | 27
  Vitality, Change at Month 6 | -6.5 (22.6)
  Vitality, Change at Month 12: number analyzed (Participants) | 22
  Vitality, Change at Month 12 | -10.2 (24.0)
  Vitality, Change at Month 24: number analyzed (Participants) | 12
  Vitality, Change at Month 24 | -14.6 (22.5)
  Vitality, Change at Month 36: number analyzed (Participants) | 10
  Vitality, Change at Month 36 | -2.5 (27.5)
  Vitality, Change at Month 48: number analyzed (Participants) | 7
  Vitality, Change at Month 48 | -7.1 (23.8)
  Vitality, Change at Month 60: number analyzed (Participants) | 6
  Vitality, Change at Month 60 | -4.2 (29.2)
  General Health Perception, Change at Month 1: number analyzed (Participants) | 30
  General Health Perception, Change at Month 1 | -3.8 (19.9)
  General Health Perception, Change at Month 3: number analyzed (Participants) | 27
  General Health Perception, Change at Month 3 | 2.4 (26.1)
  General Health Perception, Change at Month 6: number analyzed (Participants) | 28
  General Health Perception, Change at Month 6 | 0 (23.5)
  General Health Perception, Change at Month 12: number analyzed (Participants) | 23
  General Health Perception, Change at Month 12 | -5.2 (31.4)
  General Health Perception, Change at Month 24: number analyzed (Participants) | 12
  General Health Perception, Change at Month 24 | -11.3 (22.2)
  General Health Perception, Change at Month 36: number analyzed (Participants) | 10
  General Health Perception, Change at Month 36 | -14.5 (24.1)
  General Health Perception, Change at Month 48: number analyzed (Participants) | 7
  General Health Perception, Change at Month 48 | -14.3 (28.9)
  General Health Perception, Change at Month 60: number analyzed (Participants) | 6
  General Health Perception, Change at Month 60 | -22.5 (33.6)

8. Secondary Outcome: Cryoablation Technical Success of the Study Cryoablation Procedure
Description: A technically successful treatment was defined by an ablation volume encompassing the tumor with at least a 5 mm margin. Technical success was calculated on a per tumor level as well as a participant level. To be considered a technical success on a participant level, all tumors treated during the baseline procedure were required to meet the technical success criteria (that is, an ablation volume encompassing the tumor with at least a 5 mm margin).
Time Frame: Up to 60 months
Population: Participants for whom cryoablation via Galil Medical Cryoablation System was attempted or performed (ITT Population).
Measure: Number; unit: percentage of tumors
Units Other Than Participants: Tumors
Arm/Group | Cryoablation
Number analyzed (Participants) | 40
Number analyzed (Tumors) | 60
percentage of tumors | 100

9. Secondary Outcome: Number of Participants With an Intra- or Post-operative Adverse Event (AE), a Serious AE, or an Unanticipated Adverse Device Effect (UADE)
Description: An AE was defined as any untoward medical occurrence that develops or worsens in severity during the conduct of a clinical study. Serious AEs include death, a life-threatening AE, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, or an important medical event that jeopardized the participant and required medical intervention to prevent the previously listed serious outcomes. UADE was any serious adverse effect, any life-threatening problem or death caused by or associated with a device, if it was not previously identified in nature, severity, or degree of incidence in the application; or any other unanticipated serious problem associated with a device. The AEs that are presented were considered related to the cryoablation procedure. A summary of other non-serious AEs and all serious AEs, regardless of causality is located in Reported AE section.
Time Frame: Baseline up to 30 days post-cryoablation
Population: Participants for whom cryoablation via Galil Medical Cryoablation System was attempted or performed (ITT Population).
Measure: Count of Participants; unit: Participants
Arm/Group | Cryoablation
Number analyzed (Participants) | 40
Participants
  Intra-operative nonserious AE (NSAE) | 23
  Post-operative NSAE, prior to discharge | 9
  Post-operative NSAE within 30 days of procedure | 19
  Serious AE | 6
  UADE | 0

10. Secondary Outcome: Metastatic Disease Spread as Measured by Imaging
Description: Evidence of additional metastatic disease post cryoablation procedure as measured by imaging is presented.
Time Frame: Months 3, 6, 12, 24, 36, 48, and 60
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cryoablation
Number analyzed (Participants) | 40
Participants
  Month 3: number analyzed (Participants) | 38
  Month 3 | 16
  Month 6: number analyzed (Participants) | 36
  Month 6 | 14
  Month 12: number analyzed (Participants) | 35
  Month 12 | 14
  Month 24: number analyzed (Participants) | 28
  Month 24 | 10
  Month 36: number analyzed (Participants) | 24
  Month 36 | 9
  Month 48: number analyzed (Participants) | 21
  Month 48 | 7
  Month 60: number analyzed (Participants) | 17
  Month 60 | 6

ADVERSE EVENTS:
Time Frame: Baseline up to Month 60
Description: Participants for whom cryoablation via Galil Medical Cryoablation System was attempted or performed (ITT Population).
Arm/Group | Cryoablation
All-Cause Mortality (participants affected / at risk) | 20/40
Serious Adverse Events (participants affected / at risk) | 6/40
Other Adverse Events (participants affected / at risk) | 32/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cryoablation (N=40)
Appendicitis (Infections and infestations) | 1
Vascular access complication (Injury, poisoning and procedural complications) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3
Bilateral subdural hematoma (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Cryoablation (N=40)
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Fever (General disorders) | 1
Flu like symptoms (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Pain (General disorders) | 1
Pain at procedure site (General disorders) | 2
Lung infection (Infections and infestations) | 1
Skin infection (Infections and infestations) | 1
Burn (Injury, poisoning and procedural complications) | 1
Intraoperative hemorrhage (Injury, poisoning and procedural complications) | 2
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 2
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1
Pain in left arm (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 1
Vaginal inflammation (Reproductive system and breast disorders) | 1/16 — This is a sex-specific adverse event that only affects female participants.
Alveolar hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 11
Pleural hemorrhage (Respiratory, thoracic and mediastinal disorders) | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 19
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
BTG can require Investigator to postpone publications/presentations for up to 12 months so data from all sites can be published. BTG will limit review of Investigator's draft to confirm Confidential Information is not being disclosed. If BTG notes publishing Study results may affect obtaining a patent, Investigator will not publish for up to 60 days until patent application is filed. Investigator will acknowledge BTG in any publication/presentation.

DOCUMENTS (2):
  • Study Protocol (2011-08-09): https://cdn.clinicaltrials.gov/large-docs/01/NCT01307501/Prot_000.pdf
  • Statistical Analysis Plan (2012-08-27): https://cdn.clinicaltrials.gov/large-docs/01/NCT01307501/SAP_001.pdf